CLINICAL TRIAL: NCT05479461
Title: A Two-arm Parallel Randomized Clinical Trial of Implementation of Technology-enabled Management Versus Usual Care for Blood Pressure
Brief Title: Technology-enabled Management Versus Usual Care for Blood Pressure
Acronym: HrtEx
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Paul Wang, Professor of Medicine (Cardiovascular Medicine), Stanford University Medical Center, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 63700
Record Dates: First submitted 2022-07-20; First posted 2022-07-29 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Hypertension
Keywords: High blood pressure; Digital Health Mobile Technology; Cardiovascular risk; Clinical Research; Medications
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Randomized open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mobile Health Technology (Experimental)
  Interventions: Other: Digital Hypertension Management System
- Usual Care (Active Comparator)
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Digital Hypertension Management System — Mobile health technology using physician- directed, semi-automated management of hypertension
  Arms: Mobile Health Technology
Other: Usual Care — The participants will receive usual care
  Arms: Usual Care

SUMMARY:
Two arm parallel randomized clinical trial

DETAILED DESCRIPTION:
For this study, we have 3 cohorts that employ varying recruitment strategies before they are enrolled in the interventions.

At Stanford, we have 2 cohorts, where Cohort 1 is recruiting participants through clinic screening and contacting them through text or email.

For Cohort 2, recruitment is divided into two phases: Control Phase I and Intervention Phase II. During Control Phase I, standard recruitment methods were employed, including general outreach through participating clinics and pre-existing clinical networks. These efforts did not incorporate specific strategies aimed at enhancing diversity or prioritizing underrepresented populations. In contrast, Intervention Phase II introduced four targeted strategies designed to improve the inclusion of African-American, Hispanic/Latinx individuals, and women.

1. Digital Outreach via BuildClinical: The study leverages a digital recruitment campaign managed by BuildClinical, utilizing targeted online advertisements across various platforms. Prospective participants who engage with the advertisements are directed to a study landing page, where they receive detailed study information and complete a preliminary eligibility screening before being contacted by the study team.
2. Patient Registry-Based Recruitment: Eligible participants will be identified through structured data queries from the STAnford Research Repository (STARR) or EPIC registry. This approach ensures targeted outreach to individuals who meet the study's inclusion criteria while reducing screening burden.
3. Honest Broker Outreach via Stanford RPEP: To maintain privacy compliance, the Stanford Research Participant Engagement Program (RPEP) will conduct Honest Broker outreach via multiple channels, including secure Epic MyHealth messages, postal mail, and provider co-invitations. This method allows potential participants to opt in or out before direct contact with the research team, ensuring ethical and efficient recruitment.
4. Spanish-Speaking Ambassador Program: A dedicated Spanish-speaking ambassador will support recruitment efforts by engaging with Spanish-speaking participants, providing culturally tailored study information, and assisting with the informed consent process. This initiative ensures equitable access for Spanish-speaking individuals and facilitates participation among historically underrepresented populations.

   Our TIDE site partners at the Morehouse School of Medicine utilize their own recruitment methods for cohort 3, which uses the following:

   Medical residents will be randomized into three screening groups using a block randomization approach to ensure demographic balance across the groups (e.g., age, years in training, prior experience). Each group will utilize a different screening method for patient recruitment:

   Arm 1: Resident-Led Manual Screening

   Residents apply eligibility criteria manually by reviewing patient EMRs and making judgment-based decisions.

   Arm 2: AI-Assisted Screening

   AI software, Deep 6, will scan EMRs for inclusion criteria and flag potentially eligible patients. Residents will then validate flagged cases to confirm or deny eligibility.

   Arm 3: Coordinator-Led Screening (Control)

   Coordinators screen patients independently of AI, applying eligibility criteria consistently across all patient records.

   These comprehensive recruitment strategies are designed to enhance enrollment diversity, improve participant engagement, and ensure a balanced distribution of participants across study arms.

   Primary and Secondary Endpoints for Cohort 1

   Primary Endpoint
   * Percentage of participants who consent to participate following text message compared to the percentage of participants who consent to participate following emailoutreach.

   Secondary Endpoints

   ● Percentage of participants who consent following either text message or telephone outreach.

   ● Percentage of participants who consent after opting out after receiving a call or text message.
   * Median time from call/text initiation to participant response among all participants who are contacted and respond.
   * Percentage of African American, Hispanic, or Asian participants who consent to participate following text message compared to the percentage of African American, Hispanic, and Asian participants who consent to participate following email outreach.
   * Percentage of African American or Hispanic participants who consent to participate following text message compared to the percentage of African American or Hispanic, participants who consent to participate following email outreach.
   * Percentage of Asian participants who consent to participate following text message compared to the percentage of Asian participants who consent to participate following email outreach.

   Primary and Secondary Endpoints for Cohort 2

   Primary Endpoint

   ● Percentage of participants enrolled who are either African-American or Hispanic/LatinX during Intervention Phase II compared to Control Phase I.

   Secondary Endpoints

   ● Percentage of African-American or Hispanic/LatinX participants who screen positive during Intervention Phase II compared to Control Phase I.

   ● Percentage of Hispanic/LatinX participants enrolled during Intervention Phase II compared to Control Phase I.

   ● Percentage of African-American participants enrolled during Intervention Phase II compared to Control Phase I.

   ● Percentage of women participants enrolled during Intervention Phase II compared to Control Phase I.

   ● Percentage of African-American, Hispanic/LatinX, or women participants enrolled during Intervention Phase II compared to Control Phase I.

   ● Percentage of African-American, Hispanic/LatinX, or women participants who screen positive during Intervention Phase II compared to Control Phase I.

   ● Percentage of Hispanic/LatinX participants who screen positive during Intervention Phase II compared to Control Phase I.

   ● Percentage of African-American participants who screen positive during Intervention Phase II compared to Control Phase I.

   ● Percentage of women participants who screen positive during Intervention Phase II compared to Control Phase I.

   ● Percentage of African-American or Hispanic/LatinX participants contacted through Honest Broker and enrolled during Intervention Phase II compared to the Percentage of African-American or Hispanic/LatinX participants in Control Phase I.

   ● Percentage of women participants contacted through Honest Broker and enrolled during Intervention Phase II compared to the percentage of women participants in Control Phase I.

   ● Percentage of African-American or Hispanic/LatinX participants contacted through Patient Registry and enrolled during Intervention Phase II compared to the Percentage of African-American or Hispanic/LatinX participants in Control Phase I.

   ● Percentage of women participants contacted through Patient Registry and enrolled during Intervention Phase II compared to the percentage of women in Control Phase I.
   * Percentage of African-American or Hispanic/LatinX participants contacted through BuildClinical and enrolled during Intervention Phase II compared to the Percentage of African-American or Hispanic/LatinX participants contacted in Control Phase I.
   * Percentage of women participants contacted through BuildClinical and enrolled during Intervention Phase II compared to Percentage of women participants enrolled in Control Phase I.
   * Percentage of Hispanic/LatinX participants contacted through Lay Coordinator and enrolled during Intervention Phase II compared to the Percentage of African-American or Hispanic/LatinX participants contacted in Control Phase I.

   Primary and Secondary Endpoints for Cohort 3

   Primary Endpoint ● Screening Accuracy: Accuracy metrics include true positive, true negative, false positive, and false negative rates across the three arms, providing insight into each method's reliability and potential for error.

   Secondary Endpoints ● Representativeness: This measures the number and characteristics (e.g., age, race/ethnicity) of patients recruited in each arm, allowing for assessment of demographic representativeness.

   ● Enrollment Screening Efficiency: This is measured as the average time per screened patient across the three arms. Efficiency will be assessed based on total time to screen each patient from record access to eligibility determination.
   * Workload and Satisfaction: Surveys will capture resident and coordinator perceptions of workload, satisfaction, and feasibility of each method, with Likert scales and qualitative feedback (Ellis & Kasperbauer, 2020).

   Statistical Analysis Plan (SAP) Cohort 1 Analysis Methods

   The proportion of participants who consent following text message or email-telephoneoutreach will be calculated. Median and interquartile range will be estimated for the time from email /text initiation to participant response.

   Cohort 2 Analysis Methods This study aims to increase recruitment through a two-phase trial that will compare a combination of recruitment strategies through 3 distinct cohort-based recruitment strategies to assess their effectiveness to improve participant diversity and engagement. Participants are control phase I or intervention phase II.

   The primary statistical test will be a two-sample Z-test for proportions, comparing enrollment percentages in African American/Black and Hispanic/Latino between the control phase I and intervention phase II. The same method will be applied to the secondary endpoints, comparing recruitment rates across demographic subgroups and different recruitment strategies. All tests will be one-sided with α=0.05.

   Based on the preliminary data from February 2025, the control phase enrolled 135 participants, with the following distributions:
   * African American/Black: 8 (5.92%)
   * Hispanic/Latino: 17 (12.6%)

   The intervention phase II aims for a 50% increase in African American/Black and Hispanic/Latino enrollment. With a total of 270 participants (135 per phase), the power calculation indicates that the statistical power to detect this significant increase is 100%.

   Cohort 3 Analysis Methods This cohort will evaluate the efficiency, accuracy, satisfaction, and representativeness across the three screening arms. The primary metric for assessing efficiency will be the mean screening time per patient. A one-way ANOVA will be conducted to compare mean screening times among the arms, followed by post-hoc tests if significant overall differences are detected. For accuracy, the analysis will be based on true and false positive/negative rates across screening methods. Chi-square tests will be used for categorical comparisons, and logistic regression will be applied to control for potential confounding variables, such as resident training level and experience. Representativeness and satisfaction will be evaluated through the analysis of demographic characteristics, including age, race, and gender along with responses to surveys assessing workload and satisfaction. Chi-square tests will be used to analyze categorical demographic data, while the Kurskal-Wallis test will be employed to compare non-parametric Likert-scale responses across all study arms. Additionally, open-ended feedback will be thematically analyzed to enrich the interpretation of quantitative findings.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-90 yrs.
* Smartphone ownership
* Office SBP: ≥ 140 mm Hg
* ≤ 2 current anti-HTN meds
* Able to add or dose-increase at least 2 of the following classes of medications: ACE-I/ARB, diuretic, calcium channel blocker, beta-blocker, mineralocorticoid receptor antagonists (i.e., at least 2 classes are available for addition or dose- increases after excluding intolerant medications and medications currently at maximum dose)
* English or Spanish-speakers

Exclusion Criteria:

* Heart failure with reduced ejection fraction (EF < 40%)
* ESRD (GFR <15)
* Renal replacement therapy
* Pregnant
* Myocardial infarction or stroke within preceding 6 months
* Hospitalization for hypertensive emergency or malignant hypertension within preceding 6 months
* Prior solid organ transplantation
* At the clinical discretion of the investigators
* Enrolled in another clinical study

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Defined Daily Dose (DDD) | Visit 1 (Baseline), Visit-3 (6 Month follow up)
  Change in defined daily dose (DDD)

SECONDARY OUTCOMES:
Systolic Blood Pressure (SBP) | Visit-1 (Baseline), Visit-3 (6 Month follow up)
  Change in home SBP
Diastolic blood pressure (DBP) | Visit-1 (Baseline), Visit-3 (6 Month follow up)
  Change in home diastolic blood pressure (DBP)
Antihypertensive Drugs | Visit-1 (Baseline), Visit-3 (6 Month follow up)
  Change in number of antihypertensive drugs
Systolic Blood Pressure (SBP) | Visit-1 (Baseline), Visit -2 (3 Month follow up)
  Change in home SBP
Physician Survey | Visit 1 (Baseline), Visit-3 (6 Month follow up)
  Change in Survey score in Likert scale: Hypertension care and satisfaction
Clinician inertia | Visit 1 (Baseline), Visit-3 (6 Month follow up)
  Proportion of visits with blood pressure above 130/80 mm Hg where medication was not intensified

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Wang, MD, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - Stanford Health Care, Palo Alto, California
  - Morehouse School of Medicine, Atlanta, Georgia
  - Lake Country Medical Group, Eatonton, Georgia

IPD SHARING:
Plan to Share IPD: No